CLINICAL TRIAL: NCT00046904
Title: Phase III Placebo-Controlled, Randomized, Double-Blind Comparison Of Etanercept (Enbrel) Versus Placebo For The Treatment Of Cancer-Associated Weight Loss And Anorexia
Brief Title: Etanercept in Treating Cancer-Related Cachexia and Anorexia in Patients With Advanced Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Aminah Jatoi, M.D., Mayo Clinic Cancer Center
Allocation: Randomized | Masking: Double | Purpose: Supportive Care
Other Study IDs: CDR0000257027; NCCTG-N00C1; NCI-P02-0232; MC00C8 (Other: Mayo Clinic Cancer Center); 1497-00 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Last update posted 2011-05-05 (Estimated); Status verified 2011-05

CONDITIONS: Anorexia; Cachexia; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; anorexia; cachexia
MeSH Terms: conditions — Anorexia; Cachexia | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: etanercept

SUMMARY:
RATIONALE: Etanercept is a substance that is being studied as a treatment for cachexia (weight loss) and anorexia (lack of appetite) in patients who have cancer. It is not yet known whether etanercept is effective in improving cancer-related cachexia and anorexia.

PURPOSE: Randomized phase III trial to determine the effectiveness of etanercept in treating cancer-related cachexia and anorexia in patients who have advanced cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare etanercept vs placebo in the treatment of cancer-related cachexia and anorexia, in terms of weight measurement and rate of weight change, in patients with advanced malignancies.
* Determine the effect of this drug on nausea and vomiting in these patients.
* Assess the functional status and appetite of patients treated with this drug.
* Assess the quality of life of patients treated with this drug.
* Determine the toxic effects of this drug in these patients.
* Determine whether this drug prolongs survival of these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to primary malignant disease (lung vs gastrointestinal vs other), severity of weight loss (less than 4.6 kg vs at least 4.6 kg), planned concurrent chemotherapy (yes vs no), age (less than 50 vs 50 and over), gender, planned use of megestrol or other progestational agent (yes vs no), and GBU Prognostic Index (good vs bad vs unsure). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive etanercept subcutaneously (SC) twice weekly.
* Arm II: Patients receive placebo SC twice weekly. Treatment in both arms continues for a maximum of 24 weeks in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, weekly for 1 month, and then monthly during treatment.

Patients are followed every 6 months for 5 years.

PROJECTED ACCRUAL: A total of 274 patients (137 per treatment arm) will be accrued for this study within 19 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed malignancy except brain cancer

  * If the patient has multiple primaries or an unknown primary, the currently active cancer cannot be brain cancer
* Disease considered incurable with available therapies
* No clinical evidence of ascites
* Weight loss of at least 5 pounds (2.3 kg) within the past 2 months (excluding perioperative weight loss) and/or estimated caloric intake of less than 20 cal/kg daily
* Weight gain determined by physician to be beneficial
* Patient perceives weight loss as a problem

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* More than 3 months

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Cardiovascular

* No poorly controlled congestive heart failure
* No poorly controlled hypertension
* No pacemaker, implanted defibrillator, stents, or metal suture material in the heart or great vessels (for patients participating in the BIA translational portion of the study)

Gastrointestinal

* No known mechanical obstruction of the alimentary tract
* No malabsorption
* No intractable vomiting (more than 5 episodes/week)
* Not concurrently receiving tube feedings or parenteral nutrition

Other

* Able to reliably administer subcutaneous medication twice weekly
* Alert and mentally competent
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 1 month since prior infliximab
* No concurrent live vaccination

Chemotherapy

* Concurrent chemotherapy allowed

Endocrine therapy

* At least 1 month since prior adrenal steroids
* No concurrent adrenal steroids (inhalant, topical, or optical steroids allowed)

  * Concurrent short-term dexamethasone for chemotherapy-induced emesis is allowed

Radiotherapy

* Concurrent radiotherapy allowed

Surgery

* Not specified

Other

* More than 1 month since prior etanercept
* No concurrent evaluation with another device that injects an electrical current into the body (for patients participating in the bioelectrical impendance analysis [BIA] translational portion of the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-05; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Comparison of weight gain and rate of weight change

SECONDARY OUTCOMES:
Differences in appetite
Overall survival
Incidence of treatment-related toxicity
Comparison of quality of life (QOL) as assessed by the QOL UNISCALE and the Functional Assessment of Cancer Therapy-Anorexia/cachexia (FACT-An) scale at baseline, weekly for one month, and then monthly during study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, MD, Study Chair — Mayo Clinic
Locations (19):
- United States (19):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates at June E. Nylen Cancer Center, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Cancer Care Center at Medcenter One Hospital, Bismarck, North Dakota
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota

REFERENCES:
- [Result] Jatoi A, Dakhil SR, Nguyen PL, Sloan JA, Kugler JW, Rowland KM Jr, Soori GS, Wender DB, Fitch TR, Novotny PJ, Loprinzi CL. A placebo-controlled double blind trial of etanercept for the cancer anorexia/weight loss syndrome: results from N00C1 from the North Central Cancer Treatment Group. Cancer. 2007 Sep 15;110(6):1396-403. doi: 10.1002/cncr.22944. PMID 17674351
- [Result] Jatoi A, Dakhil SR, Kugler JW, et al.: A placebo-controlled trial of etanercept, a tumor necrosis factor (TNF) inhibitor, in patients with the cancer anorexia/weight loss syndrome. North Central Cancer Treatment Group (NCCTG) trial N00C1. [Abstract] J Clin Oncol 24 (Suppl 18): A-8534, 476s, 2006.